CLINICAL TRIAL: NCT00292266
Title: An Open Label, Randomized, Multicenter, Comparative, Parallel Group Study of Rebif® 44 Mcg Administered Three Times Per Week by Subcutaneous Injection, Compared With Avonex® 30 Mcg Administered Once Per Week by Intramuscular Injection in the Treatment of Relapsing-remitting Multiple Sclerosis
Brief Title: A Study of Rebif® Compared With Avonex® in the Treatment of Relapsing-remitting Multiple Sclerosis (MS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21125
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing-remitting Multiple Sclerosis; Rebif®; Avonex®; interferon-beta-1a
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

ARMS (2):
- Rebif® (Experimental)
  Interventions: Drug: Rebif®
- Avonex® (Active Comparator)
  Interventions: Drug: Avonex®

INTERVENTIONS:
Drug: Rebif® — Rebif® injection will be administered subcutaneously at a dose of 44 mcg, three times per week, up to 72 weeks.
  Arms: Rebif®
Drug: Avonex® — Avonex® injection will be administered intramuscularly at a dose of 30 mcg, once weekly, up to 72 weeks.
  Arms: Avonex®

SUMMARY:
This is an open-label, randomized, multicenter, comparative, and parallel-group study comparing the therapeutic effects of two interferon-beta-1a regimens in relapsing-remitting multiple sclerosis (MS). The primary objective is to demonstrate the superiority of Rebif® 44 microgram (mcg) subcutaneous injection given three times a week (132 mcg per week) to that of Avonex® 30 mcg intramuscular injection given once a week.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Clinically definite or laboratory-supported definite relapsing-remitting MS according to Poser's criteria
* Two or more relapses within the preceding 24 months
* Clinical stability or improving neurological state during the 4 weeks before Study Day 1
* Expanded disability status scale (EDSS) score from 0 to 5.5, inclusive
* Two or more lesions consistent with MS on a Screening proton density/T2-magnetic resonance imaging (MRI) scan to be performed 28 plus/minus (+/-) 4 days before the Study Day 1 MRI
* Willingness and ability to comply with the protocol for the duration of the study
* Written informed consent given before any study-related procedure not part of the subject's normal medical care, with the understanding that the subject can withdraw consent at any time without prejudice to future medical care
* For female subjects, lack of childbearing potential must be satisfied by either being post-menopausal or surgically sterilized or using a hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study. Subjects should neither be pregnant nor breast-feeding; confirmation that the subject is not pregnant will be established by a negative serum human chorionic gonadotropin (hCG) pregnancy test within 7 days of Study Day 1 (the pregnancy test will not be required of subjects who will be post-menopausal or surgically sterilized)

Exclusion Criteria:

* Secondary progressive MS, primary progressive MS or progressive relapsing MS
* Prior use of interferon
* Treatment with oral or systemic corticosteroids or adrenocorticotropic hormone (ACTH) within 4 weeks of Study Day 1 or within 7 days before the Screening MRI
* Psychiatric disorder that is unstable or will preclude safe participation in the study
* Significant leucopenia (white blood cell count less than 0.5 times the lower limit of normal) within 7 days of Study Day 1
* Elevated liver function tests (Alanine transaminase [ALT], Aspartate transaminase [AST], alkaline phosphatase or total bilirubin greater than 2 times the upper limit of normal) within 7 days of Study Day 1
* Prior cytokine or anti-cytokine therapy or glatiramer acetate within the 3 months before Study Day 1
* Immunomodulatory or immunosuppressive therapy within the 12 months before Study Day 1, including but not limited to cyclophosphamide, cyclosporin, methotrexate, azathioprine, linomide and mitoxantrone
* Previous use of cladribine or total lymphoid irradiation
* Allergy to human serum albumin, mannitol or gadolinium diethylenetriaminepentacetic acid (DTPA)
* Intravenous immunoglobulin or any other investigational drug or procedure in the 6 months before Study Day 1
* Systemic disease that can interfere with subject safety, compliance or evaluation of the condition under study, such as insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease or infection with human immunodeficiency virus (HIV) or Human T-cell lymphotrophic virus, Type-1 (HTLV-1)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 677 (Actual)
Dates: Start 1999-11; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Percentage of exacerbation-free subjects | Week 24
Percentage of exacerbation-free subjects | Week 48
Percentage of exacerbation-free subjects | Week 72

SECONDARY OUTCOMES:
Mean number of combined unique (CU) active lesions per subject per scan | Week 24
Total exacerbation count per subject | Week 24, 48 and 72
Mean Number of Time constant 2 (T2) active lesions per subject per scan | Week 24, 48 and 72

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Francis, M.D., Study Director — Merck Serono International SA

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com